CLINICAL TRIAL: NCT07130474
Title: Role of Long Noncoding RNA LINC01134 in Metastasis of Hepatitis C Virus-related Hepatocellular Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Elsayed Hassan, Demonstrator, Sohag University
Other Study IDs: Soh-Med-25-7-14MS
Record Dates: First submitted 2025-08-08; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: diagnosed cases of HCC without metastasis
- controls: diagnosed cases of HCC with metastasis

SUMMARY:
LINC01134, a novel lncRNA, has received increasing attention in cancer research, particularly in hepatocellular carcinoma (HCC). It had been shown that LINC01134 promotes HCC progression by facilitating tumor proliferation, migration, epithelial-mesenchymal transition, oxaliplatin resistance, and radio resistance (Wang et al,2021).

Functional experiments revealed that ectopic expression of LINC01134 promotes HCC cell migration and invasion in vitro and HCC liver metastasis and lung metastasis in vivo. Knockdown of LINC01134 represses HCC cell migration and invasion in vitro and HCC liver metastasis and lung metastasis in vivo (Wang et al, 2020).

Metastasis and recurrence are the main causes of HCC-induced deaths even with curative resection (Huang et al., 2019; Sakamoto et al., 2019). Therefore, we focused on the lncRNAs implicated in the metastasis and recurrence of HCC. In the current research, we attempted to examine the expression profile and explore the function of LINC01134 in the metastasis of HCC. It has been well established that lncRNAs expressed in the cytoplasm can serve as competitive endogenous RNAs (ceRNAs) to sponge miRNAs, by which they negatively regulate the translation of mRNAs.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCV infection will be based on positive HCV antibodies by enzyme-linked immunosorbent assay (ELISA) & HCV RNA by polymerase chain reaction (PCR) for more than 6 months. The diagnosis of liver cirrhosis will be based on clinical data and findings on abdominal ultrasound. The diagnosis of HCC will be based on the typical features of dynamic imaging by triphasic CT with or without elevated serum alpha-fetoprotein (AFP) levels (Murakami et al., 2002).

Exclusion Criteria:

* Co-infection with HBV.

  * Presence of clinically suspected other causes of hepatocellular injury (any history of alcoholism, autoimmune hepatitis, primary sclerosing cholangitis (PSC), primary biliary cholangitis (PBC), Wilson's disease, fatty liver disease with metabolic syndrome & drug-induced liver disease.
  * Patients diagnosed with other malignancies.
  * Patients with a history of prior local or systemic HCC-specific treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with hcc
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
mechanism of action of LINC01134 in metastasis of HCC via miRNA-4784/ Akt signal pathway. | -Data will be collected over 3 months.

IPD SHARING:
Plan to Share IPD: Undecided